CLINICAL TRIAL: NCT06912880
Title: Effects Of Surgical and Medical Therapy on Psychosocial, Quality Of Life and Social Participation in Women With Stress Urinary Incontinence
Brief Title: Effects of Therapies in Women With Stress Urinary Incontinence
Status: Completed | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Burçin Uğur Tosun, Principal Investigator, Eastern Mediterranean University
Other Study IDs: November 10,2017
Record Dates: First submitted 2022-07-01; First posted 2025-04-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Stress Urinary Incontinence
Keywords: quality of life; social participation; women; incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the medical treatment group: 16 female Stress Urinary Incontinence patients considered for medical treatment as anticholinergic combinations their doctors and met the inclusion criteria of the study were assessed immediately before the treatment and 8 weeks after their medical treatment. The subjects in the medical treatment group received medication procedure. All patient assessments were performed face to face by the same physiotherapist.
- the surgical treatment group: In the surgical treatment group 16 female Stress Urinary Incontinence patients underwent the Transobturator Tape (TOT) procedure. All patient assessments were performed face to face by the same physiotherapist.
  Interventions: Procedure: trans obturator tape surgery

INTERVENTIONS:
Procedure: trans obturator tape surgery — Trans-obturator technique is a more beneficial and a less invasive procedure in treatment of SUI when compared with other techiniques. In this technique, a synthetic mesh tape, which is passing bilaterally through the obturator foramen, is placed underneath the mid part of the urethra.
  Groups: the surgical treatment group

SUMMARY:
Purpose:

This study aims to evaluate how surgical and medical treatments affect quality of life, depression status, and social participation in women with stress urinary incontinence (SUI).

Methods:

The study includes 32 women diagnosed with SUI. Participants are divided into two groups: 16 receiving medical treatment and 16 undergoing surgical treatment. All participants are evaluated before treatment and 8 weeks after its completion using the following instruments: International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF), Incontinence Quality of Life Questionnaire (I-QOL), World Health Organization Quality of Life Instrument-Short Form (WHOQOL-BREF), Beck Depression Inventory (BDI), and Social Participation Questionnaire (SPQ).

DETAILED DESCRIPTION:
This study was approved by the Çukurova University Institute of Health Sciences Non-Interventional Clinical Studies Ethics Committee (Meeting no. 70, November 10, 2017, File no. 29). All procedures were conducted in accordance with the Declaration of Helsinki. Written and verbal informed consent was obtained from all participants after explaining the study's purpose and procedures.

Sample size was calculated using G*Power 3.1 software (Universität Düsseldorf, Germany). Based on previous literature, the sample was powered to detect a within-group change on the Incontinence Quality of Life Questionnaire (I-QOL), with at least 16 participants required per group to achieve 80% power and a 95% confidence interval. Necessary permissions were obtained from the hospital's urology outpatient clinic prior to data collection.

A total of 32 women over the age of 18, newly diagnosed with stress urinary incontinence (SUI) and with symptoms lasting for more than 6 months, were included. Exclusion criteria included: history of vaginal or pelvic surgery within the past 6 months, current or recurrent urinary tract infections (more than 3 in the last year), neurological or neuromuscular disease (e.g., cerebrovascular accident, Alzheimer's disease, spinal cord injury, or dementia), kidney or liver failure, illiteracy, or inability to participate in evaluations or communication.

Participants were assigned to treatment by their physicians, either medical (n=16) or surgical (n=16). The medical group received pharmacological treatment, while the surgical group underwent the Transobturator Tape (TOT) procedure. Evaluations were conducted face-to-face by the same physiotherapist before treatment and 8 weeks after treatment using standardized questionnaires: ICIQ-SF, I-QOL, WHOQOL-BREF, BDI, and SPQ.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with Stress Urinary Incontinence
* had symptoms ongoing for over 6 months.

Exclusion Criteria:

* Cases were excluded if the individual had a vaginal or pelvic operation in the last 6 months,
* an active urinary tract infection or more than 3 urinary tract infections in the past year
* a neurological or neuromuscular disease (cerebrovascular accident, Alzheimer's, spinal cord injury, or dementia), kidney or liver failure, or was illiterate or in a condition to prevent evaluation or communication.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with diagnoses of stress urinary incontinence.
Study Population: A total of 32 female patients over the age of 18, who were newly diagnosed with SUI and had symptoms ongoing for over 6 months were included in the study. Cases were excluded if the individual had a vaginal or pelvic operation in the last 6 months, an active urinary tract infection or more than 3 urinary tract infections in the past year, a neurological or neuromuscular disease (cerebrovascular accident, Alzheimer's, spinal cord injury, or dementia), kidney or liver failure, or was illiterate or in a condition to prevent evaluation or communication.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Disease-Specific Quality of Life Score (I-QOL) | Change from Baseline (Week 0) to Post-treatment (Week 8)
  Disease-specific quality of life will be assessed using the Incontinence Quality of Life Questionnaire (I-QOL). This is a 22-item questionnaire scored on a 5-point Likert scale. Scores range from 0 to 100, with higher scores indicating better quality of life.
Change in General Quality of Life Score (WHOQOL-BREF) | Change from Baseline (Week 0) to Post-treatment (Week 8)
  General quality of life will be evaluated using the World Health Organization Quality of Life Instrument - Short Form (WHOQOL-BREF). The WHOQOL-BREF includes 26 items across four domains: physical, psychological, social, and environmental. Each domain is scored separately, with scores ranging from 0 to 100, where higher scores indicate better perceived quality of life.
depression | At the beginning and at the end of 8 weeks
  Evaluation of Depression: Depression levels will be measured using the Beck Depression Inventory, a 21-item self-report instrument. Total scores range from 0 to 63, with higher scores indicating more severe depressive symptoms.
community participation | At the beginning and at the end of 8 weeks
  Evaluation of Community Participation: The Social Participation Questionnaire was used to assess the extent the subjects actively took part in life activities and how active they were. The Social Participation Questionnaire consists of 15 items. Community participation will be evaluated using the Social Participation Questionnaire (SPQ), which includes 15 items covering domains such as home and family life, social activities, and work. Scores range from 0 to 90, with higher scores indicating greater levels of social participation.

CONTACTS AND LOCATIONS:
Overall Officials: Berkiye Kırmızıgil, Asst. Prof., Study Chair — Eastern Mediterranean University
Locations (1):
- Adana State Hospital, Adana, Çukurova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided